CLINICAL TRIAL: NCT01288274
Title: Safety and Feasibility of Community Based DMPA Provision in Tigray, Ethiopia
Brief Title: Community Based Distribution of Injectable Contraceptives in Tigray, Ethiopia
Acronym: CBDDMPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: Tigray Regional Health Bureau (Unknown); Venture Strategies for Health and Development (Other); Venture Strategies innovations (Unknown)
Responsible Party: Ndola Prata, Scientific Director, Bixby Center, University of California, Berkeley
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Bixby 001
Record Dates: First submitted 2011-01-31; First posted 2011-02-02 (Estimated); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Contraception; Family Planning; Task Shifting; Community Based Distribution; DMPA
Keywords: Contraception; Family planning; Task Shifting; Community based distribution; Ethiopia; DMPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Injection by Health Extension Worker (Active Comparator): Women who receive injectable contraceptive from clinic based health extension workers (HEWs) during the study period
  Interventions: Other: Community Based administration of DMPA
- Injection by Community Health Worker (Active Comparator): Women who receive injectable contraceptive through community based distributors from community based reproductive health agents (CBRHAs) during the study period
  Interventions: Other: Community Based administration of DMPA

INTERVENTIONS:
Other: Community Based administration of DMPA — Injectable contraceptive administered by clinic based health extension worker or community based reproductive health agent using same protocol to test equivalence of community based distribution to facility based distribution

SUMMARY:
The purpose of this study was to demonstrate that with appropriate training, the provision of injectable contraceptives by community based reproductive health agents (CBRHAs) does not significantly differ from low-level clinic-based providers, or health extension workers (HEWs).

DETAILED DESCRIPTION:
The overall goal of this project was to increase contraceptive prevalence and reduce the current high unmet need for family planning in rural areas of Ethiopia. In addition, the project was intended to provide evidence to policy makers to expand community based distribution (CBD) of the injectible contraceptive, depot medroxyprogesterone acetate (DMPA), in both Tigray and other regions of Ethiopia where community based reproductive health agents (CBRHAs) or other community health workers (CHWs) are present.

Following from that, the specific aims of this project were to:

* Provide evidence that CBRHAs can safely and effectively distribute and facilitate supply of DMPA to rural women
* Demonstrate that CBRHAs can deliver DMPA with the same safety, effectiveness, and acceptability outcomes as HEWs
* Increase access to DMPA by using CBRHAs

ELIGIBILITY:
Inclusion Criteria:

* All adult women of reproductive age who approached a provider for a contraceptive method and wished to use DMPA were recruited to participate in the study
* Medically eligible to use injectable contraceptives

Exclusion Criteria:

* Health problems preventing or counter-indications for use of hormonal contraceptives
* Suspicion of pregancy
* FHI validated check list of eligibility use injectable contraceptives
* Minors age <18 years old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1062 (Actual)
Dates: Start 2008-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Equivalence of injection administration | every 3 months
  Injection site morbidities, induration etc

SECONDARY OUTCOMES:
Equivalent continuation rates | Every 3 months
  Follow up injection rates at 2nd and 3rd injection.
Knowledge of side effects among clients | Every 3 months
  The clients understand the efficacy, the drug usage, side effects and recourse for care if side effects manifest at 13 week and 6 month questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ndola Prata, MD, MSc, Principal Investigator — Bixby Center, University of California, Berkeley
Locations (3):
- Ethiopia (3):
  - Kola Tembien District Health Bureau, Kola Tembien, Tigray
  - Tigray Regional Health Bureau, Mek'ele, Tigray
  - Tanqua Aberguel District Health Bureau, Tanqua Aberguel, Tigray